CLINICAL TRIAL: NCT00518297
Title: Open Label, Multiple Dose, Sequential, Drug-Drug Interaction Study to Assess the Pharmacokinetics and Safety of Atazanavir and Raltegravir Co-Administered Twice Daily in Healthy Subjects
Brief Title: DDI HV (ATV - Merck)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI424-352
Record Dates: First submitted 2007-08-17; First posted 2007-08-20 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2008-11

CONDITIONS: HIV Infections
Keywords: Antivirals / HIV
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Raltegravir
- 2 (Active Comparator)
  Interventions: Drug: Atazanavir
- 3 (Active Comparator)
  Interventions: Drug: Atazanavir + Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Tablet, Oral, 400 mg, twice daily for 5 Days
  Arms: 1
Drug: Atazanavir — Capsule, Oral, 300 mg, twice daily for 7 Days
  Other Names: Reyataz
  Arms: 2
Drug: Atazanavir + Raltegravir — Capsule/Tablet, Oral, 300/400, twice daily for 14 Days
  Other Names: Reyataz
  Arms: 3

SUMMARY:
The purpose of this study is to to assess the effect of ATV 300 mg BID on the PK of raltegravir 400 mg BID, to assess the effect of raltegravir 400 mg BID on the PK of ATV 300 mg BID, and to assess the ECG effects of ATV 300 mg BID over 21 days, given with or without raltegravir 400 mg BID.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages of 18 to 45 years old with a body mass index (BMI) of 18 to 32 kg/m²
* Prior to enrollment, subjects must have physical and laboratory test findings within normal limits, and women of childbearing potential (WOCBP) must have a negative pregnancy test

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations.
* Use of any prescription drugs or over-the-counter acid controllers within 4 weeks prior to study drug administration
* Use of any other drugs, including over-the-counter medications and herbal preparations within 1 week prior to study drug administration

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety Assessments | Screening, Days -1, 1, 5, 6, 8, 10, 12, 13, 15, 19, 22, 26, and Study Discharge
Pharmacokinetic Assessments | Days 5, 12, and 26

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol-Myers Squibb Clinical Pharmacology Unit, Hamilton, New Jersey, United States